CLINICAL TRIAL: NCT04375579
Title: Multi-domain Assessment and Quality of Life in Patients Older Than 60 Years Receiving an Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Assessment of Elderly Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: ELDERGRAF
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200084
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Stem Cell Transplant
MeSH Terms: interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comprehensive geriatric assessment (CGA) — Questionnaires on nutritional status, autonomy and quality of life

SUMMARY:
Patients older than 60 years are more and more transplanted. Comprehensive geriatric assessment (CGA) have been developed and are currently used in patients with cancer, it has been correlated with the prognosis. There is still few data in transplanted patients and the aim of this study is to assess these patients before and after transplantation in order to monitor their general health and quality of life (QOF) and correlate them to the prognostic.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or more at time of transplantation
* Patient receiving a hematopoietic stem cell allograft for myeloid hemopathy (myeloid acute leukemia, myelodysplastic syndrome, Myeloproliferative neoplasm) or for an Acute lymphoblastic leukemia
* No opposition to participate

Exclusion Criteria:

* Patient opposed to the protocol
* Vulnerable patients protected by curatorship or administrative supervision
* Patients not covered by a social security scheme

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 60 years who received an allogeneic hematopoietic stem cell transplantation HSCT
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-10-17 (Estimated)

PRIMARY OUTCOMES:
Overall survival | at one year post allogeneic hematopoietic stem cell transplantation

SECONDARY OUTCOMES:
Overall survival | at two years post allogeneic hematopoietic stem cell transplantation
Morbidity Index | at one year
Morbidity Index | at two years
Survival without disease and chronic graft-versus-host disease | at one year post allogeneic hematopoietic stem cell transplantation
Survival without disease and chronic graft-versus-host disease | at two years post allogeneic hematopoietic stem cell transplantation
Proportion of patient with Viral Reactivation | at one year
  Reactivation of cytomegalovirus (CMV) or Epstein-Barr virus (EBV) virus
Acute graft-versus-host disease | at 100 days
Chronic graft-versus-host disease | at 1 year
Chronic graft-versus-host disease | at 2 years
Incidence of relapse | at two years
Walk test | at day 100
  Walk tests measure the functional level of patients suffering from a wide range of cardiac, respiratory, neurological, and musculoskeletal conditions.
Walk test | at one year
  Walk tests measure the functional level of patients suffering from a wide range of cardiac, respiratory, neurological, and musculoskeletal conditions.
Walk test | at two years
  Walk tests measure the functional level of patients suffering from a wide range of cardiac, respiratory, neurological, and musculoskeletal conditions.
Nutritional score | at day 100
  Nutrional score will be assessed using the simple evaluation of food intake (SEFI scale). The minimum value is 0 and the maximum is 10. The highest score mean that the patient's food intake are the same as usual.
Nutritional score | at one year
  Nutrional score will be assessed using the simple evaluation of food intake (SEFI scale). The minimum value is 0 and the maximum is 10. The highest score mean that the patient's food intake are the same as usual.
Nutritional score | at two years
  Nutrional score will be assessed using the simple evaluation of food intake (SEFI scale). The minimum value is 0 and the maximum is 10. The highest score mean that the patient's food intake are the same as usual.
Karnofsky index | at day 100
  The Karnofsky index is a synthetic indicator of the overall health status measuring, on a scale from 0 (death) to 100 (full health)
Karnofsky index | at one year
  The Karnofsky index is a synthetic indicator of the overall health status measuring, on a scale from 0 (death) to 100 (full health)
Evaluation of autonomy | at one year
  Autonomy will be evaluated using ADL and IADL score. Instrumental activities of daily living - global score range from 0 to 4.
Evaluation of Quality of life | at one year
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
  EORTC QLQ-C30 Scoring Manual. Fayers PM et al. on behalf of the EORTC Quality of Life Group. EORTC, 2001. ISBN: 2-9300.
Length of hospitalisation initially | at two years
Length of hospitalisation during the first year after graft | Up to one year
Questionnaire completion rate | At 2 years
Length of pre-grafting visit | At 2 years
Length of D100 visit | At 2 years
Length of 1year visit | At 2 years
Length of 2 years visit | At 2 years

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besancon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Lyon, Lyon
  - CHU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Hopital de la Pitié Salpetrière, Paris
  - Hopital Necker, Paris
  - Hopital Saint Louis, Paris
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided